CLINICAL TRIAL: NCT04465136
Title: The Effect of Cranial Electrotherapy Stimulation as Adjunctive Therapy on Anxiety Disorder in Elderly: an Open-label, Pilot Study
Brief Title: CES in the Elderly With Generalized Anxiety Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. The results showed significant improvement after CES; 2. Run out of study grant.
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Che-Sheng Chu, Department of Psychiatry, MD, attending physician, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kaohsiung VGH
Record Dates: First submitted 2020-03-27; First posted 2020-07-09 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: CES; Anxiety Disorders and Symptoms
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Received CES intervention (Experimental): CES with the frequency of 0.5 Hertz; current of 100~600micro-ampere, for 60 minutes, everyday for 6 weeks, total 42 sessions intervention
  Interventions: Device: CES, Alpha-Stim stimulator (Electromedical Products International, Inc., Mineral Wells, Texas, USA)

INTERVENTIONS:
Device: CES, Alpha-Stim stimulator (Electromedical Products International, Inc., Mineral Wells, Texas, USA) — CES is a brain stimulation device with 2 electrodes on the bilateral earlobe. It uses Alternating current to stimulate the brain including thalamus, vagus nerve system and influence EEG and neurotransmitters like gamma-aminobutyrate. Stimulation was applied at a current intensity that can be adjusted continuously to provide between 10 and 600 micro-ampere and frequency of 0.5Hertz for 60 minutes, everyday for 6 weeks, total 42 sessions.

SUMMARY:
The study aimed to investigate whether cranial electrotherapy stimulation(CES) could benefit anxiety symptoms, depressive symptoms, quality of sleep and quality of life in elderly patients with anxiety disorder.

DETAILED DESCRIPTION:
Several studies have shown cranial electrotherapy stimulation (CES) could decrease depression and anxiety symptoms in patients with mood disorder. However, none study so far focused on the elderly population to investigate the anti-depressant and anxiolytic effect in elderly patient with anxiety disorder. Hence, this pilot study aims to assess the safety and efficacy of CES on anxiety symptoms, depressive symptoms, sleep quality and life quality in elderly patient with anxiety disorder. The study was an open-label, one arm study. The study aimed to investigate whether cranial electrotherapy stimulation(CES) could benefit anxiety symptoms, depressive symptoms, quality of sleep and quality of life in elderly patients with anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 85 years old
* Anxiety disorder confirmed by Mini-international neuropsychiatric interview (MINI)
* HAM-A score greater than 17 points
* HAM-D score lower than 17 points
* Mini-mental state examination score of 24 or more
* No psychiatric medication adjustment within 3 months.

Exclusion Criteria:

* Comorbid with another axis I psychiatric disorder, like schizophrenia, substance use disorder or other major mental illness screened by Mini-international neuropsychiatric interview (MINI)
* Contraindications for CES
* Implanted brain medical devices or mental in the head
* History of seizures
* History of intracranial neoplasm or surgery
* Severe head injuries
* Cerebrovascular diseases
* Arrhythmia or with pacemaker implantation
* Used to receive brain stimulation therapy.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
The change of objective anxiety symptom from baseline | 1.Change from baseline HAM-A score after the 4 weeks and the 6 weeks. 2.Change from baseline HAM-A score after 4 weeks (week 10) after the full CES treatment course
  evaluate the Hamilton Anxiety Rating Scale (HAM-A) for objective anxiety Each item is scored on a scale of 0 (not present) to 4(severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
The change of subjective anxiety symptom from baseline | 1. Change from baseline BAI score after the 4 weeks and the 6 weeks. 2.Change from baseline BAI score after 4 weeks (week 10) after the full CES treatment course
  evaluate the Beck anxiety inventory (BAI) for subjective anxiety The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are: 0-7: minimal anxiety; 8-15: mild anxiety; 16-25: moderate anxiety; 26-63: severe anxiety.

SECONDARY OUTCOMES:
The change of objective depressive symptom from baseline | 1. Change from baseline HAM-D score after the 4 weeks and the 6 weeks. 2.Change from baseline HAM-D score after 4 weeks (week 10) after the full CES treatment course
  Evaluate the Hamilton Depression Rating Scale (HAM-D) for objective anxiety The Ham-D is the most widely used clinician-administered depression assessment scale. The original version contains 17 items pertaining to symptoms of depression experienced over the past week. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
The change of subjective depressive symptom from baseline | 1. Change from baseline BDI-II score after the 4 weeks and the 6 weeks. 2.Change from baseline BDI-II score after 4 weeks (week 10) after the full CES treatment course
  Evaluate the Beck depression inventory-II (BDI-II) for subjective anxiety the BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original: 0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression.
The change of quality of life from baseline: Brief version of World Health Organization Quality of Life questionnaire (WHOQOL-BREF) | 1. Change from baseline WHOQOL-BREF score after the 4 weeks and the 6 weeks. 2.Change from baseline WHOQOL-BREF score after 4 weeks (week 10) after the full CES treatment course
  Evaluate the "Brief version of World Health Organization Quality of Life questionnaire - Taiwan version" for quality of life. The WHOQOL-BREF produces a quality of life profile. It is possible to derive four domain scores. Each item is weighted on a 0-4 interval scale. The WHOQOL-BREF score is then calculated by totaling the 4 domain scores. The calculation method of the scores in a certain domain is: (summation of the scores in each domain) x 4 / (number of items in a category). The adjusted scores of each domain are as low as 4 points and as high as 20 points. The overall score ranges from 16 to 80, where higher scores denote a higher life quality.
The change of quality of sleep from baseline: Pittsburgh Sleep Quality Index (PSQI) | 1. Change from baseline PSQI score after the 4 weeks and the 6 weeks. 2.Change from baseline PSQI score after 4 weeks (week 10) after the full CES treatment course
  Evaluate the Pittsburgh Sleep Quality Index (PSQI) for quality of sleep Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Che-Sheng Chu, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital., Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feusner JD, Madsen S, Moody TD, Bohon C, Hembacher E, Bookheimer SY, Bystritsky A. Effects of cranial electrotherapy stimulation on resting state brain activity. Brain Behav. 2012 May;2(3):211-20. doi: 10.1002/brb3.45. PMID 22741094
- [Background] Schroeder MJ, Barr RE. Quantitative analysis of the electroencephalogram during cranial electrotherapy stimulation. Clin Neurophysiol. 2001 Nov;112(11):2075-83. doi: 10.1016/s1388-2457(01)00657-5. PMID 11682346
- [Background] Barclay TH, Barclay RD. A clinical trial of cranial electrotherapy stimulation for anxiety and comorbid depression. J Affect Disord. 2014 Aug;164:171-7. doi: 10.1016/j.jad.2014.04.029. Epub 2014 Apr 21. PMID 24856571
- [Background] Morriss R, Xydopoulos G, Craven M, Price L, Fordham R. Clinical effectiveness and cost minimisation model of Alpha-Stim cranial electrotherapy stimulation in treatment seeking patients with moderate to severe generalised anxiety disorder. J Affect Disord. 2019 Jun 15;253:426-437. doi: 10.1016/j.jad.2019.04.020. Epub 2019 Apr 15. PMID 31103808
- [Background] Yennurajalingam S, Kang DH, Hwu WJ, Padhye NS, Masino C, Dibaj SS, Liu DD, Williams JL, Lu Z, Bruera E. Cranial Electrotherapy Stimulation for the Management of Depression, Anxiety, Sleep Disturbance, and Pain in Patients With Advanced Cancer: A Preliminary Study. J Pain Symptom Manage. 2018 Feb;55(2):198-206. doi: 10.1016/j.jpainsymman.2017.08.027. Epub 2017 Sep 21. PMID 28870799
- [Background] Shekelle P, Cook I, Miake-Lye IM, Mak S, Booth MS, Shanman R, Beroes JM. The Effectiveness and Risks of Cranial Electrical Stimulation for the Treatment of Pain, Depression, Anxiety, PTSD, and Insomnia: A Systematic Review [Internet]. Washington (DC): Department of Veterans Affairs (US); 2018 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK493132/ PMID 29630193